CLINICAL TRIAL: NCT06546982
Title: Diagnosis and Staging of Typhoid Fever Using Surface-enhanced Raman Spectroscopy Liquid Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Aachen (Other)
Collaborators: University of Agriculture Faisalabad (Unknown); Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Roger Molto Pallares, Group Leader, University Hospital, Aachen
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Typhoid Fever SERS 01
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Intervention Model Description: Spectroscopic assessment of serum samples from healthy and typhoid fever patients to identify characteristics for diagnosis and staging.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy (Experimental): The serum samples of healthy patients will be measured.
  Interventions: Diagnostic Test: Surface-enhanced Raman Spectroscopy
- Early-stage typhoid fever (Experimental): The serum samples of early-stage typhoid fever patients will be measured.
  Interventions: Diagnostic Test: Surface-enhanced Raman Spectroscopy
- Consolidated-stage typhoid fever (Experimental): The serum samples of consolidated-stage typhoid fever patients will be measured.
  Interventions: Diagnostic Test: Surface-enhanced Raman Spectroscopy

INTERVENTIONS:
Diagnostic Test: Surface-enhanced Raman Spectroscopy — The Raman spectra of patient samples will be measured in the presence of gold nanoparticles, which will enhance the spectroscopic characteristics of serum components via near-field enhancements.

SUMMARY:
The goal of this project is to adapt the gold nanoparticle-based surface-enhanced Raman spectroscopy (SERS) technology to clinical application. In this exploratory study a measurement protocol will be established to subsequently investigate whether SERS allows to diagnose patients infected with typhoid fever as well as to stage the disease.

DETAILED DESCRIPTION:
This study on the clinical application of surface-enhanced Raman spectroscopy (SERS) is composed of two parts. First, a SERS measurement protocol will be developed to enhance the interactions between gold nanoparticles and the components of the patients samples, maximizing Raman spectroscopical signatures. Given the complex composition of human blood, which encompasses numerous biological constituents, the study focuses on serum, a component obtained through centrifugation after the removal of cells and clotting factors. Fifteen spectra will be recorded per sample. The raw spectra will be post-processed, including removal of the substrate signal, baseline correction, vector normalization, and smoothing steps.

The SERS measurement protocol established in the first section will subsequently be applied to samples of healthy and typhoid fever patients. The samples from infected patients will be confirmed with the Widal test. Multivariate data analysis will be performed to identify distinctive feature characteristics in the samples that correlate to their group (healthy and infected patients), allowing patient diagnosis, as well as the severity of the infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Nishtar Medical University
* The age range of the patients was from 18 to 70 years
* Confirmed disease with the Widal test (for typhoid fever groups)

Exclusion Criteria:

* Patients with severe concurrent diseases were excluded from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
SERS measurements to differentiate between healthy and typhoid fever patients | Through study competition, up to 1 year
  SERS assessment of healthy and typhoid fever patient samples to identify unique spectroscopical characteristics to discriminate between healthy and typhoid fever patients

SECONDARY OUTCOMES:
SERS measurements to stage typhoid fever patients | Through study competition, up to 1 year
  SERS assessment of early-stage and consolidated-stage typhoid fever patient samples to identify unique spectroscopical characteristics to stage the infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Roger Molto Pallares, Aachen, Northwest, Germany

IPD SHARING:
Plan to Share IPD: No
The study results will be published in at least one scientific article.

REFERENCES:
- [Result] Ditta A, Zhang R, Nawaz H, Majeed MI, He S, Zhuang Z, Rutten S, Shahzadi A, Yaseen S, Kiessling F, Hu J, Lammers T, Pallares RM. An exploratory clinical study of the diagnosis and staging of typhoid fever using label-free surface-enhanced Raman spectroscopy liquid biopsy. Spectrochim Acta A Mol Biomol Spectrosc. 2025 May 15;333:125864. doi: 10.1016/j.saa.2025.125864. Epub 2025 Feb 4. PMID 39938329